CLINICAL TRIAL: NCT07262411
Title: Effectiveness of a Peer-based Recovery Program: A Randomized Controlled Trial
Brief Title: Peer-based Recovery Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B-ER-114-100
Record Dates: First submitted 2025-09-25; First posted 2025-12-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Mental Disorder; Recovery, Psychological
Keywords: peer; recovery program
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Grow to Recovery program-Short Version (Experimental): Participants will receive the Grow to Recovery program -Short Version, co-led by one trained peer and one trained professional.
  Interventions: Behavioral: The Grow to Recovery program-Short Version
- Control group (No Intervention): Participants in the control group receive treatment as usual.

INTERVENTIONS:
Behavioral: The Grow to Recovery program-Short Version — The program is based on "Pathways to Recovery: A Strengths Recovery Self-help Workbook." After completing the online leader training program, one peer and one professional will conduct a 10-week Grow to Recovery program-Short Version for people with mental illness. This program covers recovery concepts, strengths, and goal setting, which will be helpful for people in recovery.
  Arms: The Grow to Recovery program-Short Version

SUMMARY:
Recovery-oriented services are currently the mainstream in the field of mental health around the world. Peer services are an alternative service option promoted by recovery advocates. Western countries have invested abundant resources in promoting peer services and providing training for peer support workers. However, peer services in Taiwan have just started. More resources need to be added to make mental health services catch up with the world trend so that people with mental illness in Taiwan can have more choices. Hence, this study aims to investigate the effectiveness of the Grow to Recovery program-Short Version co-led by a peer.

DETAILED DESCRIPTION:
The study will verify the effectiveness of the Grow to Recovery program-Short Version co-led by a peer. Based on the results of the feasibility study, an online leader training course will be established. Peer leaders and professional leaders will be recruited to receive the training and colead the Grow to Recovery program-Short Version. A total of 120 people with mental illness will be recruited and randomly assigned to either the experimental group or the control group. The pre- and post-tests as well as follow-up data collected from participants will be used to establish the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Professionals:

  1. working in the community psychiatric rehabilitation organizations
  2. being willing to co-lead the recovery program with a peer
* Peers:

  1. having a diagnosis of mental illness over 1 year
  2. living in the community
  3. being age 18 yr or older
  4. having good communication skills
  5. being willing to co-lead the recovery program with a professional
* People with mental illness

  1. having a diagnosis of mental illness over 1 year
  2. living in the community and receiving psychiatric rehabilitation services
  3. being age 18 yr or older
  4. filling out the scales independently
  5. being able to participate in a recovery group and follow the group rules

Exclusion Criteria:

* People with mental illness 1. attending another recovery-related group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Stages of Recovery Scale, SRS | Changes from Baseline at 10 weeks and 34 weeks.
  The Stages of Recovery Scale (SRS) consists of 45 items, with six subscales: the sense of hope, disability management/taking responsibility, regaining autonomy, social functioning/role performance, overall well-being, and willingness to help. A higher score means better recovery status.
General Self-Efficacy Scale, GSES | Changes from Baseline at 10 weeks and 34 weeks.
  The General Self-Efficacy Scale (GSES) contains 10 items. The GSES is rated on a four-point Likert scale, with total scores ranging from 10 to 40. A higher score means better self-efficacy.
Medical Outcomes Study Social Support Survey, MOS-SS | Changes from Baseline at 10 weeks and 34 weeks.
  The Medical Outcomes Study Social Support Survey (MOS-SS) is a multidimensional, self-administered instrument that addresses all five functions of an interpersonal relationship to assess the various functional dimensions of social support, including emotional , informational, tangible, affectionate, and positive interaction. A higher score means better social support.
The Hope Scale, THS | Changes from Baseline at 10 weeks and 34 weeks.
  The Hope Scale (THS) measures the level of sense of hope. The scale consists of 12 items, including four agency items, four pathway items, and four distracters. The THS is rated on an eight-point Likert scale, with total scores ranging from 8 to 64. A higher score means a higher sense of hope.
Taiwanese Depression Questionnaire, TDQ | Changes from Baseline at 10 weeks and 34 weeks.
  The Taiwanese Depression Questionnaire (TDQ) consists of 18 items and measures depressive conditions. The TDQ is rated on a four-point Likert scale, with total scores ranging from 0 to 54. A higher score means a more depressed mood.
Social Functioning Scale, SFS | Changes from Baseline at 10 weeks and 34 weeks.
  The Social Functioning Scale (SFS) has 36 items. A higher score means better social functioning.
Perceived Psychiatric Stigma Scale, PPSS | Changes from Baseline at 10 weeks and 34 weeks.
  The Perceived Psychiatric Stigma Scale (PPSS) measures self-stigma and has 25 items. A higher score means more severe stigma.

OTHER OUTCOMES:
Course questionnaire | Changes from Baseline at the 10th week.
  The course questionnaire aims to collect course feedback from participants. The questionnaire includes a course-satisfactory survey and open questions. A higher score means higher satisfaction.
Qualitative data | at the end of the intervention (the 10th week).
  The discussion about course feedback in the 10th class will be recorded and transcribed.
Qualitative data | Immediately after the intervention
  The researchers will conduct focus groups with peer and professional leaders of the intervention group after completing the Grow to Recovery program-Short Version. Those qualitative data will be recorded, transcribed, and analyzed.
Qualitative interview | at the 34th week
  Around 16 participants of the intervention group will have an interview after 6 months (the 34th week). The data will be recorded, transcribed, and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ching Chang, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan